

Title: Specified drug-use survey of Lotriga Granular Capsules: OCEAN3 (Outcome prevention on Cardiovascular Events by Antihyperlipidemic therapy with N3-fatty acid in Japan)

NCT Number: NCT02285166

Statistical analysis plan Approve Date: 20-AUG-2020

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

# Proofeth of Lakeder, for non-commercial use only and subject to the applicable Temes of Use

### **Table of Contents**

| 1. | 0 1 | Definitions of Terms | 1 |
|---|---|---|---|
| 1 | 1.1 | Definition | |
| 1 | 1.2 | Number of digits displayed | 3 |
| 1 | 1.3 | Significance level, confidence coefficient | .(3) |
| 1 | 1.4 | Handing of assessment period data. | 3 |
| 2.0 | | Special Drug Use Surveillance | 5 |
| 12 | 2.1 | Disposition of Subjects (Composition of subject population) Patient demographics Description of treatment (status of Lotriga treatment) | 5 |
| 2 | 2.2 | Patient demographics | 6 |
| 2 | 2.3 | Description of treatment (status of Lotriga treatment) | 9 |
| 2 | 2.4 | Description of treatment (status of statin treatment) | . 10 |
| 2 | 2.5 | Description of treatment (status of EPA product treatment) | . 10 |
| 2 | 2.6 | Description of treatment (status of active vitamin D treatment) | 11 |
| 2 | 2.7 | Pregnancy during the observation period | 11 |
| 2 | 2.8 | Treatment status of dietary therapy, exercise therapy, OTC or supplement use, and concomi | tant |
| I | medic | cations other than statins and EPA products | . 12 |
| 2 | 2.9 | | |
| 12 | 2.10 | Analysis of secondary outcome measures | |
| 2 | 2.11 | Analysis of other outcome measures | . 15 |
| 2 | 2.12 | Supplemental analysis of primary outcome measures | |
| 3.0 | | Safety analysis | . 19 |
| | 3.1 | Listing of Occurrence of Adverse Reactions and Infections in Postmarketing Surveillance, Etc. (Attac | |
| I | Form | 15) | . 19 |
| 4.0 | | Summary of the subjects in the postmarketing surveillance, etc. | . 20 |
| 4 | 4.1 | Summary of Subjects in Postmarketing Surveillance, Etc. (Attached Form 16) | . 20 |
| | | Summary of Subjects in Postmarketing Surveillance, Etc. (Attached Form 16) | |
| | | To. | |
| | , < | | |
| , 0 | 5 | | |
| KKI | | | |
| 08 | | | |
| Sico | | | |
| 100 | | | |

### 1.0 Definitions of Terms

### 1.1 Definition

| Term | Definition |
|---|---|
| Lotriga | Lotriga Granular Capsules |
| SOC | MedDRA/J System Organ Class |
| HLGT | MedDRA/J High Level Group Term |
| PT | MedDRA/J Preferred Term |
| LLT | MedDRA/J Lowest Level Term |
| Enrolled patient | Patient whose enrollment as a subject was approved |
| Subject with electronic questionnaire collected | An enrolled patient for whom an electronic questionnaire was sent by |
| Subject with electronic questionnaire not collected | An enrolled patient who is not a subject with electronic questionnaire collected |
| Locked subject | A subject with electronic questionnaire collected for whom the questionnaire |
| | completion date was entered in the PMS system and the status of the |
| | questionnaire is "Final Approval" |
| Non-locked subject | A subject with electronic questionnaire collected who is not a locked subject |
| Enrolled subject | A locked subject enrolled as a patient administered Lotriga at time of |
| administered Lotriga | enrollment |
| Enrolled subject not | A locked subject enrolled as a patient not administered Lotriga at time of |
| administered Lotriga | enrollment |
| Patient not administered | A locked subject not administered Lotriga |
| Lotriga | |
| Patient administered | A locked subject who is not a patient not administered Lotriga |
| Lotriga | |
| Safety-evaluable subject | A locked subject included as a safety-evaluable subject, i.e., a subject to whom |
| 100 | none of the following apply |
| ₹0, | Treated before the contract period |
| 79. | Enrolled 15 or more days after prescribing Lotriga |
| rec | No data after start of observation |
| Safety-evaluable subject | Not administered Lotriga |
| Safety-unevaluable subject | A locked subject excluded from the safety analysis set |
| Efficacy-evaluable subject | A locked subject included as efficacy-evaluable, i.e., a subject who has no |
| | major protocol violations, is evaluable for efficacy, and none of the following |
| | apply |
| | Not on a statin |
| | Does not have hyperlipidemia |
| Efficacy-unevaluable | A locked subject excluded from the efficacy analysis set |
| Primary prevention subject | An efficacy-evaluable subject who is not a secondary prevention subject |

| | Term | Definition |
|---|---|---|
| | Secondary prevention | An efficacy-evaluable subject who meets any of the following conditions |
| | subject | Has the risk factor "history of myocardial infarction or angina |
| | | pectoris." |
| | | Has a history of PCI/CABG |
| | Age | If observation start month and day < birthday, calculated as observation start |
| | | year - birth year - 1 |
| | | If observation start month and day ≥ birthday, calculated as observation start |
| | | year - birth year |
| | | If day of birth is unknown, calculated as 1st day of the month. |
| | BMI | Calculated as Body weight (kg) / (0.0001 x Height (cm)) x Height (cm)). |
| | | Displayed to 1 decimal place, rounding off the second decimal place. |
| | Observation start date | In patients administered Lotriga, treatment start date. In patients not |
| | | administered Lotriga, patient enrollment date |
| | Observation end date | The last day of observation |
| | Observation period (days) | The total observation period. The first and last day of the observation period |
| | | are the same as "observation start date" and "observation end date," |
| | | respectively. Calculated as Observation end date - Observation start date +1. |
| | Duration of treatment | The total period of time that Lotriga is administered. The total of each duration |
| | (days) | of Lotriga treatment recorded on the questionnaire. (The total number of days |
| | | that the drug was actually administered, excluding times off the drug) |
| | | Calculated as Treatment end date - Treatment start date + 1 for each duration |
| | | of treatment. |
| | Mean daily dose | Calculated as Daily dose x Total duration of treatment at each dose / |
| | | Observation period. See above for calculation of observation period. |
| | LDL cholesterol | Blood will be drawn for the laboratory test when the subject is fasting. |
| | (Friedewald formula) | Triglycerides will be calculated with the following equation if less than |
| | (mg/dL) | 400mg/dL. Displayed as an integer only, rounding off the first decimal place. |
| | 20. | Total cholesterol - HDL cholesterol - Triglycerides / 5 |
| | 1600 | Note that LDL cholesterol is not calculated if "Total cholesterol - HDL |
| | ( 3/C | cholesterol - Triglycerides / 5" ≤ 0. |
| S | non-HDL cholesterol | Blood will be drawn for the laboratory test after a meal. Triglycerides will be |
| 4 | (mg/dL) | calculated with the following equation if $\geq$ 400mg/dL. Displayed as an integer |
| 'd' | | only, rounding off the first decimal place. |
| | | Total cholesterol - HDL cholesterol |
| | TC / HDL-C ratio | Calculated with the following equation. Displayed to 1 decimal place, |
| | | rounding off the second decimal place. |
| | | Total cholesterol / HDL cholesterol |

| Term | Definition |
|---|---|
| LDL-C / HDL-C ratio | Calculated with the following equation. Displayed to 1 decimal place, |
| | rounding off the second decimal place. |
| | LDL cholesterol (Friedewald formula) / HDL cholesterol |
| PCI | Percutaneous coronary intervention |
| CABG | Coronary artery bypass grafting |
| TG | Triglycerides |
| Summary statistics | Number of subjects, mean, standard deviation, minimum, first quartile, |
| | median, third quartile, maximum |

### 1.2 Number of digits displayed

| Term | Definition |
|---|---|
| Summary statistics | Mean: |
| | Displayed to one place of the source data, rounding off the second place of |
| | the source data. |
| | Standard deviation: |
| | Displayed to two places of the source data, rounding off the third place of the |
| | source data. |
| | First quartile, median, third quartile: |
| | Displayed to one place of the source data, rounding off the second place of |
| | the source data. |
| | Minimum, maximum: |
| | The same number of places as the source is displayed. |
| Confidence interval | Displayed to two places of the source data, rounding off the third place of the |
| | source data. |
| P value | Displayed to 4 decimal places, rounding off the fifth place. |
| 100 | If less than 0.0001, displayed as "<.0001." |

### 1.3 Significance level, confidence coefficient

Significance level: 5% (two-sided test)

Confidence coefficient 95% (two-sided estimation)

### 1.4 Handing of assessment period data

Assessment periods are defined as start of observation, 6, 12, 18, 24, 30, and 36 months after start of observation, and last assessment time point.

In the case of multiple data for a particular period, the absolute value of the difference in the number of days from the basis number of days will be calculated and the date with the smallest absolute value will be used for that assessment period. If the absolute value is the same, the latter date of testing or measurement will be used. The last assessment time point is defined as the value tested or measured on the latest date within the period of 1170 days from the observation start date (including values tested or measured during off-drug periods). In counting the number of days elapsed from the observation start date, the observation start date is defined as Day 0 and the previous day as Day -1.

| Assessment period | Time window (Number of days from the observation start date) | Basis Number of<br>Days |
|---|---|---|
| Start of observation | -90 to 0 | 0 |
| 6 months after start of observation | 1 to 270 | 180 |
| 12 months after start of observation | 271 to 450 | 360 |
| 18 months after start of observation | 451 to 630 | 540 |
| 24 months after start of observation | 631 to 810 | 7200 |
| 30 months after start of observation | 811 to 990 | 900 |
| 36 months after start of observation | 991 to 1170 | 1080 |
| Last assessment time point | 1 to 1170 | _ |
| 36 months after start of observation Last assessment time point Last assessment time point | 55° | |

### 2.0 Special Drug Use Surveillance

<Lotriga Granular Capsules [OCEAN3]>

2.1 Disposition of Subjects (Composition of subject population)

| 1 Disposition of Subjects (Composition of subject population) | |
|---|---|
| Subjects tabulated Enrolled patients in relevant Special Drug Use Surveillance | |
| for analysis | |
| Information | Number of enrolled patients, number of study sites with enrolled patients, number of |
| tabulated for | subjects with electronic questionnaire collected, number of subjects with electronic |
| analysis | questionnaire not collected, number of locked subjects, number of non-locked |
| | subjects, number of enrolled subjects administered Lotriga, number of enrolled |
| | subjects not administered Lotriga, number of safety-evaluable subjects, number of |
| | safety-unevaluable subjects, number of efficacy-evaluable subjects, and number of |
| | efficacy-unevaluable subjects |
| | A site where subjects are enrolled in different departments should not be counted |
| | more than once in the number of study sites with enrolled patients. |
| | For subjects with electronic questionnaires not collected, the number of subjects with |
| | electronic questionnaires not collected for each of the following reasons and total |
| | number of subjects |
| | <reason collecting="" for="" not="" questionnaire=""></reason> |
| | Survey in progress |
| | Questionnaire could not be collected |
| | - Investigator moved |
| | Due to the health of the investigator |
| | Enrolled 15 or more days after prescribing Lotriga (before collection |
| | of electronic questionnaire) |
| | Other |
| ~ | For safety- and efficacy-unevaluable subjects, number of subjects excluded for each |
| of l | of the following reasons and total number of subjects. If multiple reasons apply to |
| syeda. Fo | the same subject, the subject will be tabulated more than once. |
| 90. | <reasons analysis="" exclusion="" for="" from="" safety="" set=""></reasons> |
| yes. | Treated before the contract period |
| Y.o | Enrolled 15 or more days after prescribing Lotriga |
| | No data after start of observation |
| | Not administered Lotriga |
| | <reasons analysis="" efficacy="" exclusion="" for="" from="" set=""></reasons> |
| | Non-target disease |
| | Exclusion criteria violation |
| | Items for which the number of subjects is 0 are not to be output. |
| | A listing with the reasons for exclusion will be prepared for safety- and efficacy- |

| | unevaluable subjects. |
|------------------|-----------------------|
| Figure and Table | Figure 2.1, Table 2.1 |
| Nos. | |

### 2.2 Patient demographics

| | .2 Fattent demographics | | |
|---|---|---|---|
| 8 | Subjects tabulated | Efficacy-evaluable subjects in relevant Special Drug Use Surveillance | |
| - | for analysis | | 101° |
| | Information | Each item will be classified by the follow | wing categories, and the number of subjects |
| | tabulated for | and frequency will be tabulated. These | e tabulations will be performed in enrolled |
| | analysis | subjects administered Lotriga, enrolled | subjects not administered Lotriga, and in a |
| | | pooled population of the two. | 2/64 |
| | | | we. |
| | | Item C | Category |
| | | Category of patient in E | Enrolled subjects administered Lotriga, |
| | | surveillance en | nrolled subjects not administered Lotriga |
| | | Sex | Male, female |
| | | Age | Summary statistics |
| | | 4.0 < | 65 years, $\geq$ 65 years to $\leq$ 75 years, $\geq$ 75 |
| | | off' ye | rears |
| | | Number of risk factors 2, | , 3, 4, 5, 6 |
| | | (Itemization) | |
| | | Hypertension A | Absent, Present |
| | | Type 2 diabetes mellitus A | Absent, Present |
| | | Chronic kidney disease A | Absent, Present |
| | | 01 | Absent, Present |
| | adai. For no | infarction or angina | |
| | (d) | pectoris | |
| | . 40 | History of cerebral A | Absent, Present |
| | 9.0. | infarction | |
| | N. | Peripheral artery disease A | Absent, Present |
| $\cap$ | | Breakdown of risk factors | |
| | | (history of myocardial infarction | |
| | | or angina pectoris) (may be | |
| | | counted more than once) | |
| | | *Only if history of myocardial | |
| | | infarction or angina pectoris M | Ayocardial infarction, angina pectoris |
| | | "present" | |
| | | Myocardial infarction / | |

| Details on history of myocardial infarction "Only if history of myocardial infarction "present" Time of onset (closest to observation start date) Number of past episodes Details on history of cerebral infarction "present" Time of onset (closest to observation start date) Number of past episodes Details on history of cerebral infarction "present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG "Only if history of PCI/CABG "Only if history of PCI/CABG "Only if history of PCI/CABG "present" Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention "Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics <25 kg/m², 25 to <30 kg/m², ≥30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost datly [≥5 days a week!) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 times every 3 months, Other | | | | 10 | |
|---|---|---|---|---|---|
| infarction *Only if history of myocardial infarction "present" Time of onset (closest to observation start date) Number of past episodes Details on history of cerebral infarction *Only if history of cerebral infarction "present" Time of onset (closest to observation start date) Number of past episodes I, 2, 3 or more Within last year, prior to last year observation start date) Number of past episodes I, 2, 3 or more Within last year, prior to last year observation start date) Number of past episodes I, 2, 3 or more Within last year, prior to last year observation start date) Number of past episodes I, 2, 3 or more Within last year, prior to last year observation start date) History of PCI/CABG Only if history of PCI/CABG "present" Time performed (closest to observation start date) Details on history of peripheral artery intervention Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | angina pectoris | |
| *Only if history of myocardial infarction "present" Time of onset (closest to observation start date) Number of past episodes Details on history of cerebral infarction "present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Only if history of PCI/CABG Only if history of PCI/CABG "present" Time performed (closest to observation start date) History of peripheral artery intervention Only if history of peripheral artery intervention Time performed (closest to observation start date) Within last year, prior to last year observation start date) Within last year, p | | | | Details on history of myocardial | |
| infarction "present" Time of onset (closest to observation start date) Number of past episodes Details on history of cerebral infarction "present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Details on history of PCI/CABG Number of past episodes History of PCI/CABG Only if history of PCI/CABG "Only if history of PCI/CABG "Present" Time performed (closest to observation start date) History of PCI/CABG "Present" Time performed (closest to observation start date) History of peripheral artery intervention "Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "Only if history of peripheral artery intervention" Time performed (closest to observation start date) BMI Summary statistics 225 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | infarction | |
| Time of onset (closest to observation start date) Number of past episodes Details on history of cerebral infarction "only if history of cerebral infarction present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Only if history of PCI/CABG "Only if history of PCI/CABG "present" Time performed (closest to observation start date) History of PCI/CABG "present" Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention "Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to <30 kg/m², ≥30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | *Only if history of myocardial | |
| observation start date) Number of past episodes Details on history of cerebral infarction "Only if history of cerebral infarction "present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Only if history of PCI/CABG "Only if history of PCI/CABG "Only if history of PCI/CABG "present" Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention Tonly if history of peripheral artery intervention Only if history of peripheral artery intervention Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily ≥ 5 days a week ) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | infarction "present" | |
| Details on history of cerebral infarction "Only if history of cerebral infarction "Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Details on history of PCI/CABG "Only if history of PCI/CABG "Only if history of PCI/CABG "Only if history of PCI/CABG "present" Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily ≥ 5 days a week ) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | Time of onset (closest to | Within last year, prior to last year |
| infarction "present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Details on history of PCI/CABG "Only if history of PCI/CABG "Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m². Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | observation start date) | .< |
| infarction "present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Details on history of PCI/CABG "Only if history of PCI/CABG "Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m². Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | Number of past episodes | 1, 2, 3 or more |
| infarction "present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Details on history of PCI/CABG "Only if history of PCI/CABG "Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m². Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | Details on history of cerebral | 2/6 |
| infarction "present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Details on history of PCI/CABG "Only if history of PCI/CABG "Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m². Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | infarction | : Cal |
| infarction "present" Time of onset (closest to observation start date) Number of past episodes History of PCI/CABG Details on history of PCI/CABG "Only if history of PCI/CABG "Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m². Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | *Only if history of cerebral | |
| observation start date) Number of past episodes History of PCL/CABG Details on history of PCL/CABG *Only if history of PCL/CABG "present" Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention *Only if history of peripheral artery intervention Only if history of peripheral artery intervention *Only if history of peripher | | | | infarction "present" | 26, |
| Number of past episodes History of PCI/CABG Details on history of PCI/CABG "only if history of PCI/CABG "present" Time performed (closest to observation start date) History of peripheral artery intervention Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | Time of onset (closest to | Within last year, prior to last year |
| History of PCI/CABG Details on history of PCI/CABG *Only if history of PCI/CABG *Only if history of PCI/CABG *Only if history of PCI/CABG *Only if history of PCI/CABG *Only if history of PCI/CABG *Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | observation start date) | 10 |
| Details on history of PCI/CABG *Only if history of PCI/CABG *Only if history of PCI/CABG *present" Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | Number of past episodes | 1, 2, 3 or more |
| *Only if history of PCI/CABG "present" Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | History of PCI/CABG | Absent, Present |
| Time performed (Closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention "Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily ≥ 5 days a week]) Hospital visit frequency Within last year, prior to last year | | | | Details on history of PCI/CABG | 3 |
| Time performed (closest to observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention "Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics ⟨25 kg/m², 25 to ⟨30 kg/m², ≥30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily ≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | *Only if history of PCI/CABG | \$ |
| observation start date) History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention "Ornly if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | "present" | |
| History of peripheral artery intervention Details on history of peripheral artery intervention Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency Absent, Present Within last year, prior to last year Within last year, prior to last year Vithin last year, prior to last year | | | | Time performed (closest to | Within last year, prior to last year |
| intervention Details on history of peripheral artery intervention *Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | observation start date) | |
| Details on history of peripheral artery intervention *Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | History of peripheral artery | Absent, Present |
| artery intervention Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | intervention | |
| *Only if history of peripheral artery intervention "present" Time performed (closest to observation start date) BMI Summary statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Unknown Smoking history Never smoked, Current smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency *Only if history of peripheral artery intervention "present" Within last year, prior to last year Within last year, prior to last year Within last year, prior to last year Very statistics < 25 kg/m², 25 to < 30 kg/m², ≥ 30 kg/m², Very smoker, Very smoker, Previous smoker/current non-smoker Alcohol use (Drinks alcoholic beverages almost daily [≥ 5 days a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | Details on history of peripheral | |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | | artery intervention | |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | | ~ | *Only if history of peripheral | |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | ~9 | ) | artery intervention "present" | |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | 1.01 | | Time performed (closest to | Within last year, prior to last year |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | · · · · · | | observation start date) | |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | | 600 | | BMI | Summary statistics |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | _ | 3/2 | | | $<25~kg/m^2,25~to <30~kg/m^2, \geq 30~kg/m^2,$ |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | × | | | | Unknown |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | K | | | Smoking history | Never smoked, Current smoker, Previous |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | Seles | | | | smoker/current non-smoker |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | 2404 | | | Alcohol use (Drinks alcoholic | Yes, No |
| a week]) Hospital visit frequency ≥ Twice a month, About once a month, 1-2 | X | | | beverages almost daily [ $\geq 5$ days | |
| | | | | a week]) | |
| times every 3 months, Other | | | | Hospital visit frequency | ≥ Twice a month, About once a month, 1-2 |
| | | | | | times every 3 months, Other |

| | | - No. of the Control | |
|---|---|---|---|
| | | Fish consumption frequency | Almost every day, About once every 2 days, |
| | | | Once-twice a week, Almost never, Missing |
| | | | data |
| | | Previous or concurrent cerebral | Absent, Present |
| | | or cardiac vascular disorders | |
| | | Details on previous or | |
| | | concurrent cerebral or cardiac | 25 |
| | | vascular disorders | <0° |
| | | *Only if previous or concurrent | |
| | | cerebral or cardiac vascular | 630 |
| | | disorders "present" | olio |
| | | (Itemization) | 201 |
| | | Atrial fibrillation | we. |
| | | Left ventricular | Absent, Present |
| | | hypertrophy | C. C. |
| | | Cardiac failure | Absent, Present |
| | | Cerebral hemorrhage | Absent, Present |
| | | Subarachnoid hemorrhage | Absent, Present |
| | | Transient ischemic attack | Absent, Present |
| | | (TIA) | Absent, Present |
| | | Aortic aneurysm | Absent, Present |
| | | Aortic dissection | Absent, Present |
| | | Details on previous or | |
| | | concurrent cerebral hemorrhage | |
| | | *Only if prayious or conguerant | |
| | | cerebral hemorrhage "present" | |
| | 20 | Time of onset (closest to | Within last year, prior to last year |
| | of I. | observation start date) | - |
| | . 40 | Number of past episodes | 1, 2, 3 or more |
| | 98. | Details on previous or | |
| | 2/4° | concurrent subarachnoid | |
| ξ. | | hemorrhage | |
| 10 | | *Only if previous or concurrent | |
| O'KO | | subarachnoid hemorrhage | |
| -106 | akedai. Foi no | "present" | |
| 8, | | Time of onset (closest to | Within last year, prior to last year |
| | | observation start date) | |
| | | Number of past episodes | 1, 2, 3 or more |
| | | Family history of coronary artery | Absent, Present |

| | disorders (parents, siblings) | |
|---|---|---|
| | Family history of cerebrovascular disorders (parents, siblings) | Absent, Present |
| | TG (mg/dL) within 3 months | Summary statistics |
| | before start of observation (Start | < 200 mg/dL, ≥ 200 mg/dL |
| | of observation) | |
| Figure and Table | Table 2.2 | 70 |
| Nos. | | |

### 2.3 Description of treatment (status of Lotriga treatment)

| 2 | bescription of the | uu | ient (status of Louiga treatment) | 0. |
|---|---|---|---|---|
| | Subjects tabulated | Ef | fficacy-evaluable subjects in relevan | nt Special Drug Use Surveillance |
| | for analysis | | | **0 |
| | Information | Ea | ach item will be classified by the fo | llowing categories, and the number of subjects |
| | tabulated for | ar | nd frequency will be tabulated. The | ese tabulations will be performed in a pooled |
| | analysis | po | opulation of enrolled subjects adr | ninistered Lotriga and enrolled subjects not |
| | | ad | Iministered Lotriga. | |
| | | 1 | Item | Category |
| | | | Lotriga treatment (during the | Absent, Present |
| | | | observation period) | |
| | | | Details of Lotriga treatment | |
| | | | *Only if Lotriga treatment | |
| | | | "present" | |
| | | 6 | Starting dose | 2 g, 4 g, other |
| | 10 | | Change in daily dose | Absent, Present |
| | ₹0. | | Description of change in | |
| | 79. | | daily dose | $< 2 \text{ g}, 2 \text{ to} < 4 \text{ g}, 4 \text{ to} < 6 \text{ g}, \ge 6 \text{ g}$ |
| | Tec | | Mean daily dose | 1 to 30 days, 31 to 90 days, 91 to 180 days, |
| | (Q) | | | 181 to 360 days, 361 to 720 days, 721 to |
| ,0 | | | Duration of treatment | 1080 days, ≥ 1081 days |
| CHIS | Figure and Table Nos. | Т | able 2.3 | |
| .000 | Nos | 10 | 2.3 | |
| )( | 1103. | _ | | |

### 2.4 Description of treatment (status of statin treatment)

| Subjects tabulated | Efficacy-evaluable subjects in relevant Special Drug Use Surveillance | |
|---|---|---|
| for analysis | | |
| Information | Each item will be classified by the fo | llowing categories, and the number of subjects |
| tabulated for | and frequency will be tabulated. Th | ese tabulations will be performed in enrolled |
| analysis | subjects administered Lotriga, enroll | ed subjects not administered Lotriga, and in |
| | pooled population of the two. | 101 |
| | | 2/8 |
| | Item | Category |
| | Statin treatment | Absent, Present |
| | Details of statin treatment | 26, |
| | *Only if statin treatment | "HE |
| | "present" | *0 |
| | Type (may be counted more | Pravastatin sodium, simvastatin, fluvastatin |
| | than once) | sodium, atorvastatin calcium, pitavastatin |
| | | calcium, rosuvastatin calcium |
| | 20 | |
| | ONINO | |
| | Duration of treatment | 1 to 30 days, 31 to 90 days, 91 to 180 days, |
| | (during observation period) | 181 to 360 days, 361 to 720 days, 721 to |
| | ,0,0 | 1080 days, ≥ 1081 days |
| Figure and Table | Table 2.4 | |
| Nos. | offi, | |

### 2.5 Description of treatment (status of EPA product treatment)

| Subjects tabulated | Efficacy-evaluable subjects in relevant Special Drug Use Surveillance |
|---|---|
| for analysis | |

| Information | | Each item will be classified by the following categories, and the number of subjects | |
|---|---|---|---|
| tabulated | for | and frequency will be tabulated. These tabulations will be performed in enrolled | |
| analysis | | subjects administered Lotriga, enroll | ed subjects not administered Lotriga, and in a |
| | | pooled population of the two. | |
| | | Item | Category |
| | | EPA product treatment | Absent, Present |
| | | Details of EPA treatment | |
| | | *Only if EPA product treatment | 200 |
| | | "present" | ::Cal |
| | | Reason for treatment (may | Lipid control, occurrence of cardiovascular |
| | | be counted more than once) | event (or increased risk thereof), request of |
| | | | patient, other |
| Figure and | Table | Table 2.5 | 1,0 |
| Nos. | | | · eC |

## 2.6 Description of treatment (status of active vitamin D treatment)

| | | | ¥ |
|---|---|---|---|
| | Subjects tabulated | Efficacy-evaluable subjects in relevant Special Drug Use Surveillance | |
| | for analysis | OUI), | |
| | Information | Each item will be classified by the fo | llowing categories, and the number of subjects |
| | tabulated for | and frequency will be tabulated. Th | ese tabulations will be performed in enrolled |
| | analysis | subjects administered Lotriga, enroll | ed subjects not administered Lotriga, and in a |
| | | pooled population of the two. | |
| | | alul. | |
| | | Item | Category |
| | ~ | Active vitamin D treatment | Absent, Present |
| | Figure and Table | Table 2.6 | |
| | Nos. | | |
| | 169.0 | | |
| 2.7 | Pregnancy during | the observation period | |
| Oroperty of | Subjects tabulated | Safety-evaluable women who receive | red Lotriga in the relevant Special Drug Use |
| CHA | for analysis | Surveillance | |
| .08 | | | |
| Pro | | | |
| ×20 | | | |

| Subjects tabulated | Safety-evaluable women who received Lotriga in the relevant Special Drug Use |
|---|---|
| for analysis | Surveillance |

| Information | Each item will be classified by the following categories, and the number of subjects | |
|---|---|---|
| tabulated for | and frequency will be tabulated. | |
| analysis | | |
| | Item | Category |
| | Presence/absence of pregnancy | Absent, Present |
| | during the observation period | |
| | | 173 |
| Figure and Table | Table 2.7 | 70 |
| Nos. | | 2/6 |

2.8 Treatment status of dietary therapy, exercise therapy, OTC or supplement use, and concomitant medications other than statins and EPA products

| inculcations on | ici man statins and EFA products | 0. |
|---|---|---|
| Subjects tabulated | Efficacy-evaluable subjects in relevant Special | Drug Use Surveillance |
| for analysis | , *\O | |
| Information | Each item will be classified by the following categories, and the number of subjects | |
| tabulated for | and frequency will be tabulated for each asse | ssment period. These tabulations will |
| analysis | be performed in enrolled subjects administ | ered Lotriga, enrolled subjects not |
| | administered Lotriga, and in a pooled populati | on of the two. The tabulations will be |
| | based on the assessment time points on the que | estionnaire. |
| | However, any data at 12 months after start of | observation or at discontinuation will |
| | be handled as data at 6 months if there is no da | ata at 6 months and will be handled as |
| | data at 12 months if there is data at 6 months. I | n the same manner, data at 36 months |
| | after start of observation or at discontinuation | of observation will be handled as data |
| | at 18 months if there is no data at 18 months an | d will be handled as data at 24 months |
| | if there is data at 18 months. Further, data from | 24, 30, and 36 months will be handled |
| | in the same manner. | |
| " C | | |
| akedai. For no | Item | Category |
| · a· | Presence or absence of dietary therapy | Absent, Present |
| 1000 | Presence or absence of exercise therapy | Absent, Present |
| 3/2 | Use of OTC or supplements | Absent, Present, Unknown |
| | (Breakdown for "present"; may be | |
| | counted more than once) | EPA, DHA, vitamin D, other |
| | Administration of hyperlipidemia | Absent, Present |
| | treatment (other than statins, Lotriga, or | |
| | EPA) | |
| | (Breakdown for "present"; may be | Anion exchange resin, small |
| | counted more than once) | intestinal cholesterol transporter |

| | | nicotinic acid products, other |
|---|---|---|
| | Administration of antihypertensives | Absent, Present |
| | (Breakdown for "present"; may be | ARB, ACE-I, CCB, α-blockers, β- |
| | counted more than once) | blockers, αβ-blockers, diuretics, |
| | | renin inhibitors, other |
| | Administration of antidiabetics | Absent, Present |
| | (Breakdown for "present"; may be | SUs, BG agents, α-GIs, TZDs, |
| | counted more than once) | DPP-4 inhibitors, GLP-1 receptor |
| | | agonists, SGLT-2 inhibitors, |
| | | glinides, insulin products, other |
| | Administration of antiplatelet drugs | Absent, Present |
| | (Breakdown for "present"; may be | Aspirin, ticlopidine, clopidogrel, |
| | counted more than once) | cilostazol, other |
| | Administration of anticoagulants | Absent, Present |
| | (Breakdown for "present"; may be | Warfarin, factor Xa inhibitors, |
| | counted more than once) | thrombin inhibitors, other |
| | Administration of nitrates | Absent, Present |
| Figure and Table | Table 2.8 | • |
| Nos. | · H | |

| | Nos. | |
|---|---|---|
| 2.0 | 2.9 Analysis of primary outcome measures | |
| 2.9 | The state of the s | ( 0 |
| | Subjects tabulated | Efficacy-evaluable subjects in relevant Special Drug Use Surveillance |
| | for analysis | |
| | Information | [Analysis of primary outcome measures] |
| | tabulated for | First onset of any of the following cardiovascular events |
| | analysis | The following key major cardiovascular events |
| | 'akeda: For no | Major cardiovascular event |
| | 10, | 1) Cardiovascular death (sudden death, fatal myocardial infarction, fatal |
| | ý. | cardiac failure, fatal stroke [cerebral infarction, cerebral hemorrhage, |
| | , eou | subarachnoid hemorrhage], other cardiovascular death) |
| _ | St | 2) Non-fatal myocardial infarction |
| 3 | | 3) Non-fatal stroke (cerebral infarction, cerebral hemorrhage, |
| | | subarachnoid hemorrhage) |
| | | <ul> <li>Anginal pectoris requiring coronary revascularization (PCI or CABG)</li> </ul> |
| | | <ul> <li>Peripheral artery disease requiring surgery or peripheral artery intervention</li> </ul> |
| | | [Description of analysis] |
| | | The following analysis will be performed. If no events occur during the observation |
| | | period (the period from the observation start date to the observation end date), the |

censoring time point will be the observation period end date.

- Kaplan-Meier estimates of cumulative incidence every 6 months in enrolled subjects administered Lotriga and enrolled subjects not administered Lotriga
- II. Comparison of enrolled subjects administered Lotriga and enrolled subjects not administered Lotriga, based on a Cox proportional hazards model, using as covariates age (continuous value), sex, BMI, smoking history, fish consumption frequency, presence or absence of previous or concurrent cerebral or cardiac vascular disorders, fasting triglycerides (continuous value), presence or absence of administration of antihypertensives, presence or absence of administration of antidiabetics, presence of administration of antiplatelet drugs, presence or absence of administration of anticoagulants, and number of risk factors (continuous value).
- III. For covariates whose interactions with the treatment group are statistically significant at a significance level of 5% when a Cox proportional hazard model with all of the covariates in II., freatment group, and interactions between the covariates and the treatment group is applied to the primary endpoint, the following analyses will be performed:

Estimates of cumulative incidence by every 6 months by each category\* of the covariates by the treatment group based on Kaplan-Meier methods Comparison of the treatment group based on a Cox proportional hazard model with only the treatment group.

(\*: for the continuous covariates, the following categorization will be made. age: "<65 years,  $\geq$  65 years to < 75 years,  $\geq$  75 years," BMI: "< 25 kg/m2, 25 to < 30 kg/m2,  $\geq$  30 kg/m2," fasting triglycerides: "< 200 mg/dL,  $\geq$  200 mg/dL," and number of risk factors: "2, 3, or 4 to 6")

The level at which smoking history and fish consumption frequency are collected on the questionnaire will be changed according to the following logic.

Smoking history: "Current smoker," "previous smoker/current non-smoker," and "missing data" will be consolidated into one level.

Fish consumption frequency: Missing data will be handled as one level.

The same analysis as in III. will be performed in the respective subgroups of primary prevention subjects and secondary prevention subjects by presence or absence of history of myocardial infarction, angina pectoris, cerebral infarction, or cerebral hemorrhage and by presence or absence of history of coronary revascularization.

For reference, the same analyses as in I and II will be performed in "patients administered Lotriga and patients not administered Lotriga" instead of "enrolled subjects administered Lotriga and enrolled subjects not administered Lotriga."

Figure and Table

Table 2.9

14

| 1 |
|---|
| 1 |
| 1 |
| 1 |

### 2.10 Analysis of secondary outcome measures

| 10 Analysis of secon | dary outcome measures |
|---|---|
| Subjects tabulated | Efficacy-evaluable subjects in relevant Special Drug Use Surveillance |
| for analysis | |
| Information | [Secondary outcome measures] |
| tabulated for | [1] All deaths (cardiovascular deaths and deaths other than cardiovascular deaths) |
| analysis | [2] First onset of any of the following key major cardiovascular events |
| | [3] First onset of any of the following cardiovascular events |
| | Major cardiovascular events |
| | Cardiovascular death (sudden death, fatal myocardial infarction, fatal |
| | cardiac failure, fatal stroke [cerebral infarction, cerebral hemorrhage, |
| | subarachnoid hemorrhage], other cardiovascular death) |
| | Non-fatal myocardial infarction |
| | 3) Non-fatal stroke (cerebral infarction, cerebral hemorrhage, |
| | subarachnoid hemorrhage) |
| | Angina pectoris requiring hospitalization* |
| | <ol> <li>Anginal pectoris requiring coronary revascularization (PCI or CABG)</li> </ol> |
| | 4. Cardiac failure requiring hospitalization |
| | <ol><li>Transient ischemic attack requiring hospitalization</li></ol> |
| | <ol><li>Peripheral artery disease requiring hospitalization*</li></ol> |
| | 7. Peripheral artery disease requiring surgery or peripheral artery intervention |
| | *Including percutaneous revascularization performed on an out-patient |
| | basis. |
| | [4] Onset of individual cardiovascular events |
| ~ | [Description of analysis] |
| 1.01 | The same analysis will be performed as the analysis in I. and II. for the primary |
| | outcome measure. |
| Figure and Table | Table 2.10 |
| Nos. | |

| | | outcome measure. |
|---|---|---|
| | Figure and Table | Table 2.10 |
| | Nos. | |
| O. | | |
| 2.1 | 1 Analysis of other | outcome measures |
| property 2.1 | Subjects tabulated | Efficacy-evaluable subjects in relevant Special Drug Use Surveillance |
| 200 | for analysis | |
| Α. | Information | [Other outcome measures] |
| | tabulated for | [1] First onset of any of fatal myocardial infarction, non-fatal myocardial infarction, |
| | analysis | and angina pectoris requiring hospitalization |
| | | [2] First onset of any of fatal stroke, non-fatal stroke, and transient ischemic attack |

| each testing time point - Test value at start of observation) at each testing time point |
|---|
| outcome measure. Among the items in [3], summary statistics for test values and change (Test value for |
| The same analysis will be performed as the analysis in [1] and [2] for the primary |
| [Description of analysis] |
| electrocardiogram |
| HbA1c [NGSP value]), and occurrence of clinically significant changes in |
| HDL-C, TC/HDL-C ratio, LDL-C/HDL-C ratio, EPA, DHA, AA, DHLA, and |
| [3] Time-course of vital signs (systolic blood pressure, diastolic blood pressure, and<br>heart rate), time course of laboratory test results (TG, TC, HDL-C, LDL-C, non- |
| requiring hospitalization |

| | Nos. | 72 |
|---|---|---|
| 2.1 | , and | |
| 2.1 | | llysis of primary outcome measures |
| | Subjects tabulated | Efficacy-evaluable subjects in relevant Special Drug Use Surveillance |
| | for analysis | |
| Î | Information | [Analysis of primary outcome measures] |
| | tabulated for | First onset of any of the following cardiovascular events |
| | analysis | The following key major cardiovascular events |
| | | Major cardiovascular events |
| | | Cardiovascular death (sudden death, fatal myocardial infarction, fatal) |
| | ~9 | cardiac failure, fatal stroke [cerebral infarction, cerebral hemorrhage, |
| | 101 | subarachnoid hemorrhage], other cardiovascular death) |
| | | Non-fatal myocardial infarction |
| | akeda: For no | 3) Non-fatal stroke (cerebral infarction, cerebral hemorrhage, |
| | The state of the s | subarachnoid hemorrhage) |
| X | , , | Anginal pectoris requiring coronary revascularization (PCI or CABG) |
| 0, | | Peripheral artery disease requiring surgery or peripheral artery intervention |
| | | [Description of analysis] |
| | | The following supplemental analysis of the above primary outcome measures will be |
| | | performed using propensity scores. |
| | | The propensity scores for each subject will be estimated using a logistic regression |
| | | model in which the probability of assignment to the Lotriga treatment group |

converted to a logit is the response variable and the following items are the objective variables.

The covariates to be included in the propensity score model are defined as follows. Age (continuous value), sex, BMI, smoking history, fish consumption frequency, presence or absence of previous or concurrent cerebral or cardiac vascular disorders, fasting triglycerides (continuous value), presence or absence of administration of antihypertensives, presence or absence of administration of antidiabetics, presence or absence of administration of antiplatelet drugs, presence or absence of administration of anticoagulants, number of risk factors (continuous value)

The level at which smoking history and fish consumption frequency are collected on the questionnaire will be changed according to the following logic.

Smoking history: "Current smoker," "previous smoker/current non-smoker," and "missing data" will be consolidated into one level.

Fish consumption frequency: Missing data will be handled as one level.

[2] Weighted analysis using inverse probability weighting (IPW)\*

### [1] Distribution of propensity scores

Summary statistics will be calculated for estimated propensity scores. In addition, the number and proportion of subjects in categories produced by demarcating propensity scores by the quartiles will be tabulated. This tabulation will be performed separately from that performed by enrolled subjects administered Lotriga and enrolled subjects not administered Lotriga.

Using IPW for each subject, Kaplan-Meier estimates of cumulative incidence every 6 months in enrolled subjects administered Lotriga and enrolled subjects not administered Lotriga and Cox regression with treatment group (enrolled subjects administered Lotriga and enrolled subjects not administered Lotriga) included in the model will be performed. As necessary, logistic regression (where the model includes treatment group) and doubly robust estimation with IPW will be performed, handling events in the primary outcome measure as binary data (presence or absence of event). The explanatory variables included in the outcome regression model in the doubly robust estimation will be the same as in the propensity score model. Estimates, standard error, and twosided 95% confidence interval will be calculated for the treatment groups in the

# Property of Yakeda. For no [3] Propensity score matching

One-to-one nearest neighbor matching without replacement using 0.2-fold the standard deviation of estimated propensity scores converted to logits as the calipers will be applied. The standard difference between enrolled subjects

Cox regression, logistic regression, and doubly robust estimation. Robust

decentralization will be used for the standard error.

| | administered Lotriga and enrolled subjects not administered Lotriga will be calculated for variables used for estimating propensity scores before and after matching. In propensity-matched populations, Kaplan-Meier estimates of cumulative incidence every 6 months in enrolled subjects administered Lotriga and enrolled subjects not administered Lotriga and Cox regression analysis with treatment group (enrolled subjects administered Lotriga and enrolled subjects not administered Lotriga) included in the model will be performed. As necessary, logistic regression (where the model includes treatment group) will be performed, handling events in the primary outcome measure as binary data (presence or absence of event). Estimates, standard error, and two-sided 95% confidence interval will be calculated for the treatment groups in the Cox regression and logistic regression. Robust decentralization will be used for the standard error. [4] Weighted analysis using matching weight (MW)* The same analysis as in [2] will be performed with MW weighting for each subject. However, a bootstrap approach will be used in the doubly robust estimation. [5] Other As necessary, analysis with a marginal structural Cox model will be |
|---|---|
| F: 1.T.11 | performed using covariates, etc., estimated every 6 months. |
| Figure and Table | Table 2.12 |
| Nos. | 3). A Weighting Analogue to Pair Matching in Propensity Score Analysis. Int J Biostat, |
| 31:9(2):215-34 | 5). A weighting Analogue to Fair Matching in Propensity Score Analysis. Int 3 Biostat, |
| 31;9(2):215-34. | Sn.commi |

### 3.0 Safety analysis

3.1 Listing of Occurrence of Adverse Reactions and Infections in Postmarketing Surveillance, Etc.

### (Attached Form 15)

| Subjects tabulated | Safety-evaluable subjects in relevant Special Drug Use Surveillance | |
|---|---|---|
| for analysis | | |
| Information | The following items will be tabulated from each postmarketing surveillance, etc. | |
| tabulated for | Item | Information tabulated for analysis |
| analysis | Number of safety- | Number of subjects in the "subjects tabulated for |
| | evaluable subjects | analysis" (above) from the relevant analysis. |
| | Number of subjects with | Number of subjects who experienced adverse drug |
| | adverse drug reactions, | reactions, etc. |
| | etc. | reactions, etc. |
| | Percentage of subjects | This will be calculated as Number of subjects with |
| | with adverse drug | adverse drug reactions, etc. / Number of safety- |
| | reactions, etc. | evaluable subjects x 100. |
| | | When performing the analysis the following |
| | | method will be employed. |
| | à | [Types of adverse drug reactions, etc.] |
| | 0,0 | MedDRA/J will be used for coding adverse |
| | , USE | drug reactions, etc. Adverse drug reactions, |
| | Minercialuseon | etc., will be tabulated by SOC and then by PT |
| | eic. | within the SOCs. For the SOC of |
| | aine | "Investigations," adverse drug reactions, etc. |
| | col, | will be tabulated by HLGT (arranged in |
| | 0,7 | ascending order of HLGT codes, but not |
| 100 | Types of adverse drug | output) and then by PT. |
| 601 | reactions, etc. | The number of subjects with and incidence of |
| \$0. | | adverse drug reactions, etc. will be listed in |
| akeda. Fo | | the Internationally Agreed Order of SOCs. If |
| SIL | | the same SOC occurs multiple times in the |
| | | same subject, it will be counted as 1 subject |
| | | in that SOC. |
| | | For PTs, the number of subjects with and |
| | | incidence of adverse drug reactions, etc. will |
| | | be listed in ascending order of PT codes. If |
| | | the same PT occurs multiple times in the |
| | | same subject, it will be counted as 1 subject |
| | | with that PT. |

| Figure and Table | Table 3.1 |
|------------------|-----------|
| Nos. | |

- 4.0 Summary of the subjects in the postmarketing surveillance, etc.
  - 4.1 Summary of Subjects in Postmarketing Surveillance, Etc. (Attached Form 16)

| 10.00 | | Commence of the second of the |
|---|---|---|
| | Subjects tabulated | Subjects with collected questionnaires in relevant Special Drug Use Surveillance |
| | for analysis | X Offi |
| | Information | Listings will be prepared for the following items in accordance with (Notes 1-3) of |
| | tabulated for | Attached Form 16 in "Re-examination Notification," Notification No. 1128-2, of the |
| | analysis | Pharmaceutical Evaluation Division, PSEHB, dated November 28, 2017. |
| | | Item |
| | | Subject No. |
| | | Site |
| | | Sex |
| | | Date of birth |
| | | Reason for use (disease code, disease name) |
| | | Complications (disease code, disease name) |
| | | Route of administration |
| | | Maximum dose |
| | | Mean dose |
| | | Unit |
| | | Duration of use |
| | | Conconntant drugs (drug code, drug name) |
| | | Extent of effect |
| | | Adverse drug reactions (disease code, disease name, outcome) |
| | ~ | Questionnaire No. |
| | , of | Dropouts |
| | Figure and Table | Table 4.1 |
| | Nos O | |
| | SK | |
| S. | | |
| Property of | | |
| Self | | |
| 2504 | | |
| X | | |